CLINICAL TRIAL: NCT06235021
Title: Clinical Efficacy of Saffron Mouth Rinse in Periodontitis Patients With Renal Disease: A Randomized Controlled Clinical Trial
Brief Title: Clinical Efficacy of Saffron Mouth Rinse in Periodontitis Patients With Renal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Dalia Ghalwash, Professor, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-064
Record Dates: First submitted 2024-01-02; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Diseases; Periodontal Pocket; Periodontal Inflammation
Keywords: Saffron; Renal; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Periodontitis

STUDY DESIGN:
Intervention Model Description: The experimental group will receive scaling and root debridement and will be instructed to use a mouthwash containing aqueous extract of saffron twice a day for 6 weeks.
Who Masked: Outcomes Assessor
Masking Description: The clinical outcome assessor (A.A) will not be aware of which treatment will be being administered, thus yielding a single-blind controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saffron (Experimental): The experimental group will receive scaling and root debridement and will be instructed to use a mouthwash containing aqueous extract of saffron twice a day for 6 weeks.
  Interventions: Other: Saffron
- chlorhexidine mouthwash. (Placebo Comparator): The control group will receive scaling and root debridement and gargle their mouth with commercial product of 0.2% chlorhexidine mouthwash.
  Interventions: Other: chlorhexidine mouthwash

INTERVENTIONS:
Other: Saffron — Saffron powder (purchased from Moayeri Copmany2 in Oman, prepared from the stigma of Crocus sativus L.).
  Total of 10 mg of saffron powder will be added to 100 ml of distilled water. Then, it will be incubated on a shaker for 24 h. The material will be passed through several layers of muslin cloth. The extracts will then be poured into a round bottom balloon and placed in the freezer at a temperature of -80°C. After freezing, the extracts were placed in a freeze-dryer.
  In vacuum, the solvent will be removed and saffron powder will be obtained. After preparing the initial concentration, serial dilution with ratios of one-half and one-third will be performed in sterile vials and one-half of the final concentration will be discarded.
  After the preparation of extract, the 0.2% saffron mouthwash will be prepared by mixing the following ingredients: 1. propylene glycol (5 g) 2. saffron extract (0.2 g) 3. polysorbate 80 (1.8 g) 4. sodium benzoate (0.2 g) 5. water (91 g).
  Arms: Saffron
Other: chlorhexidine mouthwash — commercial product of 0.2% chlorhexidine mouthwash.
  Arms: chlorhexidine mouthwash.

SUMMARY:
The commensal oral bacteria are responsible for the initiation and propagation of the disease through the process of dysbiosis, or microbial imbalance. The disease proceeds cyclically with periods of activity and quiescence until therapeutic action is taken, or the tooth and surrounding structures are destroyed by the disease process that may result in the loss of the tooth. As periodontal disease progresses from gingivitis to periodontitis, a greater number of anaerobic organisms colonize deeper periodontal pockets, such as Aggregatibacter actinomycetemcomitans and Porphyromonas gingivalis, which triggers the host inflammatory response. This response includes the production and dissemination of C-reactive protein (CRP), a biomarker of inflammation, as well as various neutrophil and macrophage compounds such as tumor necrosis factor-alpha (TNF-a), matrix metalloproteinases (MMPs), and interleukins (IL-1 and IL-8). An elevated serum CRP level suggests that the inflammation arising as a result of periodontitis may correlate with cardiovascular pathology. Additionally, smoking creates an increasingly favorable environment for the growth of periodontal pathogens, thus furthering the disease process.

In recent meta-analysis, published articles on the effect of saffron supplementation on three inflammatory biomarkers (CRP, TNF-α, and IL-6) were evaluated. Combining eight eligible trials, it was demonstrated that saffron supplementation did not have a significant effect on serum levels of the three inflammatory biomarkers. However, in the subgroup analysis, saffron was found to significantly reduce CRP and TNF-α serum concentrations

DETAILED DESCRIPTION:
Periodontitis, a common inflammatory dis ease, affects the teeth-supporting tissues. In this complex disease, dental biofilm interacts with inflammatory immune system, which may lead to an imbalance between bacterial invasion and the intensity of the host immune response. Scaling and root planning (SRP) is a common major meth od used as the gold standard for periodontal treatment. However, SRP alone has limited effects on some bacterial species and does not remove subgingival bacteria completely. This may be related to the fact that some species may exist in soft tissue, dentinal tubules, or root surface irregularities, which are associated with the treatment failure.

Therefore, to help the healing process, both chemical and herbal therapeutic mouthwashes were added to the treatment. In this way, herbs such as turmeric with its potent anti-inflammatory active ingredient, curcumin, or ginger have been used as adjunctive treatment for periodontitis along with SRP. In traditional Persian medicine, saffron and its extracts are used to improve digestion, increase appetite, relaxation, and treat liver diseases, spasm, toothache, rhinitis, pharyngitis, insomnia, depression, cough, asthma, bronchitis, fever, nausea, scarlet fever, urinary tract infections, cardiovascular disorders, and even cancers and immune system modulation. According to the modern studies, saffron has antioxidant, anti-inflammatory, anticoagulant, antibacterial and analgesic effects.

In recent years, herbal plants have received increasing attention considering their roles in health and disease. Saffron (Crocus sativus, L.) is an example of herbs, commonly used as a flavoring agent in food preparation. Saffron contains high amounts of carotenoid pigments (crocin, crocetin, α-carotene, lycopene, and zeaxanthin), monoterpene aldehydes (picrocrocin and safranal), monoterpenoids (crocusatines), isophorones, and flavonoids, which could contribute to its wide range of biological properties. A number of investigations have shown that saffron possesses anti-oxidant, anti-tumor, anti-genotoxic, and hypotensive properties. In addition, a growing number of studies have suggested that saffron possesses anti-inflammatory properties too.

However, clinical studies are very limited about the use of saffron in the field of oral diseases. A laboratory study reported that ethyl acetate extract of saffron has strong antimicrobial effects against various microorganisms such as both gram-positive (g+) and gram-negative (g-) bacteria, but it is obvious that alcoholic compounds themselves may have an antibacterial effect, so to avoid errors, the investigators chose the aqueous type from two types of alcoholic and aqueous extracts.

Considering the anti-inflammatory effect of saffron and due to the dissatisfaction of some patients with the taste of conventional mouthwashes, especially the gold standard chlorhexidine, this study was conducted to investigate the effect of mouthwash containing saffron aqueous extract on periodontal indices of patients with moderate to severe generalized periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* - Both genders, aged above 18 years.
* All patients must have a periodontal disease.
* Patients must be able to make reliable decision or communications.

Exclusion Criteria:

* - Smoking, Alcohol.
* Vulnerable groups such as pregnant females, prisoners, mentally and physically handicapped individuals.
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment loss (CAL) | 6 weeks
  With a periodontal probe, pocket depth (PD) and clinical attachment loss (CAL) will be measured on six locations of the teeth (mesio-buccal/facial, mid-buccal/facial, disto-buccal/facial, mesio-lingual/palatinal, mid-lingual/palatinal, disto-lingual/palatinal).

SECONDARY OUTCOMES:
Bleeding on probing | 6 weeks
  The proportion of bleeding sites 10 second after being stimulated by a standardized manual probe with a controlled force to the bottom of the sulcus/pocket at six locations (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual) on all present teeth will be assessed dichotomously as a BOP score on all present teeth
Plaque index | 6 weeks
  An index for the entire mouth is determined by dividing the total score by the number of surfaces examined.Quigley-Hain plaque index0No plaque1Isolated flecks of plaque at the gingival margin2A continuous band of plaque up to 1mm at the gingival margin3Plaque greater than 1mm in width and covering up to one third of the tooth surface4Plaque covering from one thirds to two thirds of the tooth surface5Plaque covering more than two thirds of the tooth surface higher scores indicate worse outcome and lower scores indicate better outcome
Gingival crevicular fluid (C- reactive protein) | 6 weeks
  The gingival crevicular fluid (GCF) will collected from PPD ≥ 5 mm in control and interventional sides for each patient from two buccal sites of two different teeth GCF will be collected by using Periopaper (Oraflow Inc) strip before scaling at baseline and after 6 weeks at the same sites during the review visit.
  The collection method will adapted. Samples will be collected in the morning, between 9 am to 12.30 pm. Prior to GCF collection, supragingival plaque and calculus will be carefully removed by using a hand scaler.
  higher scores indicate worse outcome and lower scores indicate better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Ghalwash, Study Director — The British University in Egypt
Locations (1):
- The British University in Egypt, Cairo, Egypt